CLINICAL TRIAL: NCT05935722
Title: Evaluation of a Home-based Parenting Support Program - Parenting Young Children - for Parents With Intellectual and Developmental Disabilities When There is a Risk for Neglect
Brief Title: Evaluation of a Home-based Parenting Support Program: Parenting Young Children
Acronym: PYC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Linkoeping University (Other Government); Mälardalen University (Other); Stockholm University (Other); Uppsala University (Other); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORU 4.2-00340/2023
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Intellectual Disability; Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder
Keywords: Intellectual and developmental disabilities; parents; parenting skills; support programme
MeSH Terms: conditions — Intellectual Disability; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Developmental Disabilities | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenting Young Children (Experimental): Home based parenting programme for supporting parent with IDDs. 3-6 months of structured coaching sessions.
  Interventions: Behavioral: Parenting Young Children
- Treatment as Usual (Active Comparator): Variety of interventions as usually provided by the social services.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Parenting Young Children — PYC is a home-based intervention programme involving weekly, one-hour sessions over a period of at least six months. The programme has two core modules (1) Parent-Child Interaction and (2) Child Care Skills and Safety. The Parent-Child Interaction module focuses on the parent-child relationship and interaction skills such as parents' responsiveness to the child's signals, giving the child attention and encouragement, and supporting prosocial behaviour. The Child Care Skills and Safety module targets safety at home and the parent's caring skills (e.g. food, health, and hygiene). Checklists are adapted to each parent in order to support the PYC practitioner and the parent. The programme is compiled in a manual that includes work tasks, instructions for how to perform the tasks, and teaching materials.
  Arms: Parenting Young Children
Behavioral: Treatment as Usual — TAU consists of a variety of interventions from the social services. The support will be logged and classified in accordance with the Swedish National Board of Health and Welfare's guidelines for classifications of its activities. TAU will be divided into the following five categories: 1) conversation counselling or emotional support, 2) practical support, 3) skills training, 4) compensatory strategies, and 5) other support. Support will also be classified based on whether it is home-based or given outside the home and whether it is individualised or in a group setting.
  Arms: Treatment as Usual

SUMMARY:
Background: Parents with intellectual and developmental disabilities (IDDs) have a tendency to provide insufficient caregiving and often need parenting support to prevent neglect and child removal. However, parents with IDDs are not provided with appropriate support, and there is a lack of evidence-based programmes tailored to these parents' needs. Parenting Young Children (PYC) is a home-based parenting programme developed for parents with IDDs. PYC has shown promising clinical results in interview-based studies, but there is no evidence of its effectiveness. The purpose of the proposed study is to evaluate the PYC programme for improving parenting in parents with IDDs where there is risk of child neglect. The study will include a quantitative evaluation, a process evaluation, and a qualitative evaluation of the children's and parents' perspectives on participating in PYC.

Methods: The quantitative evaluation will have a multi-centre, non-randomised, comparative study design. Eligible for participation are parents with IDDs who have children aged 0-9 years living at home and who are assessed as needing tailored parenting support. Thirty parents receiving PYC and thirty parents receiving treatment as usual (TAU) will be recruited from Swedish municipal social services. Outcome variables will be examined before and after the intervention, with a follow-up 6 months after completing the intervention. The primary outcome will be goal-attainment in parenting skills, and secondary outcomes will be parental self-efficacy and children's wellbeing. Interview methods will be used to explore the perspectives of parents and children in the PYC group.

Discussion: This study is motivated by the need for evidence-based support for parents with IDDs, and it focuses on upholding the centrality of child-caregiver relationships and family preservation, as well as children's rights and the rights of people with disabilities. Social services have expressed ethical concerns with employing a randomized design for this vulnerable group, and this study will therefore evaluate PYC in a non-randomized comparative study.

ELIGIBILITY:
Inclusion Criteria:

* Parents with IDDs, including ID and other cognitive disabilities (e.g., ADHD and ASD).
* Parents must have children aged 0-9 years living at home and be assessed by the social services to be eligible for tailored parenting support.

Exclusion Criteria:

* Ongoing substance abuse, and/or mental illness of such nature and degree that it may affect parent management training.
* Ongoing child abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure, performance sub-scale. | Baseline (pre-intervention), 3-6 months (post-intervention), 9-12 months (follow-up)
  1 Item, reported as 1-10 points.
Change in Canadian Occupational Performance Measure, satisfaction sub-scale. | Baseline (pre-intervention), 3-6 months (post-intervention), 9-12 months (follow-up)
  1 Item, reported as 1-10 points.

SECONDARY OUTCOMES:
Change in Parental Sense of Competence Scale. | Baseline (pre-intervention), 3-6 months (post-intervention), 9-12 months (follow-up)
  15 items, reported as 15-90 points.
Strengths and Difficulties Questionnaire. | Baseline (pre-intervention), 3-6 months (post-intervention), 9-12 months (follow-up)
  25 items, reported as 0-50 points.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Strandberg, PhD, Principal Investigator — Örebro universitet
Locations (5):
- Sweden (5):
  - Social Welfare Office, Enköping
  - Social Welfare Office, Jönköping
  - Social Welfare Office, Motala
  - Social Welfare Office, Tierp
  - Social Welfare Office, Uppsala

IPD SHARING:
Plan to Share IPD: No